CLINICAL TRIAL: NCT02497274
Title: Obesity and Lipids: a Matter of Taste? Impact of Bariatric Surgery on Taste Receptors
Brief Title: Obesity and Lipids: a Matter of Taste?
Acronym: HumanFATaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C14-77; 2015-A00906-43 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: bariatric surgery; taste perception; lipid receptors
MeSH Terms: conditions — Obesity | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roux Y gastric bypass (Experimental): candidates for bariatric surgery by Roux Y gastric bypass with taste assessment and epithelium gustatory smear and biopsy
  Interventions: Other: taste assessment and epithelium gustatory smear and biopsy
- Sleeve gastrectomy (Experimental): candidates for bariatric surgery by sleeve gastrectomy with taste assessment and epithelium gustatory smear and biopsy
  Interventions: Other: taste assessment and epithelium gustatory smear and biopsy

INTERVENTIONS:
Other: taste assessment and epithelium gustatory smear and biopsy — assessment of taste perceptions and expression of taste receptors before and after bariatric surgery and epithelium gustatory smear and biopsy

SUMMARY:
The purpose of the protocol is to determine the impact of bariatric surgery on taste receptors and taste perceptions and to precise the factors implicated in taste alterations in 50 obese patients before and 6 months after bariatric surgery (25 Roux Y gastric bypass and 25 sleeve gastrectomy).

DETAILED DESCRIPTION:
Over-consumption high sugar and high fat foods was identified as a main risk factor for obesity. The recent identification of lipid-receptor (CD36, GPR120) in human taste buds suggests that lipids could be perceived not only by their texture and their olfactory characteristics, but also by way of taste. Obese subjects tend to consume more high fat foods than lean subjects. Conversely, bariatric surgery induces behavioral changes limiting the consumption of foods high in sugar and fat. The mechanisms underlying these behavioral changes are not understood. Does obesity is accompanied by a distortion of taste detection of dietary lipids? What are the mechanisms involved? Are they reversible? What could be the effect on food choices and health? This protocol is part of a broader research program that aims to answer these questions by studying the feeding behavior in obese subjects and animals before and after a bariatric surgery.

The purpose of the protocol is to determine the impact of bariatric surgery on the expression of taste receptors and taste perceptions and in particular the threshold of perception of fat (and sweet as taste as reference) and to study the association between the changes of taste perceptions and food preferences, amount of weight loss, surgical technique (with or without intestinal bypass), hormonal, metabolic and inflammatory changes, and modification of the oral microbiota. The study will included 50 patients who underwent bariatric surgery, either Roux Y gastric bypass (25 patients) or sleeve gastrectomy (25 patients) that will be explored in the two months before and six months after surgery. These explorations will included a clinical examination with collection of anthropometric data, a body fat determination by impedance, a detailed dietary survey, blood samples for assessment of hormonal parameters (GLP1 , PYY, ghrelin, insulin, leptin) and inflammatory parameters (LPS, TNFalpha, IL-1, IL-6, ...), a tong micro-biopsy to collect taste buds and a sample of oral microbiota and lipids and sugars thresholds determination (linoleic acid or sucrose).

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to a health insurance
* Patients candidates for bariatric surgery based on criteria established by international experts (BMI> 40 or> 35 kg / m² with severe comorbidities, after failure of multidisciplinary care for a period of at least 1 year)
* Written consent after oral and written informations

Exclusion Criteria:

* Topic guardianship, curatorship or safeguard justice.
* Taking a treatment known to alter the perception of taste
* Oral Decay can affect the perception of taste
* Treatment that may interfere with intestinal peptides or lipids receptors (especially DDP4 inhibitors, anti-inflammatory medications, intestinal lipase inhibitors: Xenical)
* Tobacco use, alcohol or drugs abuse
* Known coagulopathy, abnormal hemostasis tests or abnormal platelets count, treatment interfering with coagulation or platelet aggregation
* Contraindication to bariatric surgery
* Malignant pathology, severe liver disease or severe inflammatory disease, malabsorption.
* Pregnancy
* Positive serology for VIH, VBH and CVH

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Expression of lipid receptors | before and 6 months after bariatric surgery
  To compare the expression of lipid receptors expressed in the taste buds before and after a significant weight loss induced by bariatric surgery

SECONDARY OUTCOMES:
Lipids thresholds | before and 6 months after bariatric surgery
  To determine the relationship between taste receptor expression and changes in lipid and sugar perception thresholds before and after surgery

OTHER OUTCOMES:
Factors associated with taste perception | before and 6 months after bariatric surgery
  To identify the factors associated with the expression and functionality of taste receptors before and after bariatric surgery: body fat, metabolic, endocrine and inflammatory parameters and peripapillary microbiota.
Influence of surgical technique on taste perception | before and 6 months after bariatric surgery
  To compare the effect of RYGBP which bypass the proximal gut with changes in intestinal endocrine secretions and lipid absorption, to that of SG that is a pure restrictive technique without intestinal bypass.

CONTACTS AND LOCATIONS:
Overall Officials: Séverine Ledoux, Principal Investigator — APHP-INSERM

REFERENCES:
- [Result] Bernard A, Le Beyec-Le Bihan J, Radoi L, Coupaye M, Sami O, Casanova N, Le May C, Collet X, Delaby P, Le Bourgot C, Besnard P, Ledoux S. Orosensory Perception of Fat/Sweet Stimuli and Appetite-Regulating Peptides before and after Sleeve Gastrectomy or Gastric Bypass in Adult Women with Obesity. Nutrients. 2021 Mar 8;13(3):878. doi: 10.3390/nu13030878. PMID 33800516
- [Result] Bernard A, Richard C, Radoi L, Boidot R, Ledoux S, Besnard P. Fat taste sensitivity in women with obesity: transcriptomic analysis of fungiform papillae before and after bariatric surgery. Obesity (Silver Spring). 2025 Aug;33(8):1518-1528. doi: 10.1002/oby.24325. Epub 2025 Jun 22. PMID 40545805
- [Result] Bernard A, Radoi L, Christensen J, Servant F, Blasco-Blaque V, Ledoux S, Collet X, Besnard P. A specific tongue microbiota signature is found in patients displaying an improvement of orosensory lipid perception after a sleeve gastrectomy. Front Nutr. 2023 Jan 11;9:1046454. doi: 10.3389/fnut.2022.1046454. eCollection 2022. PMID 36712531